CLINICAL TRIAL: NCT05938426
Title: Digital Therapeutics (ET-101) Research on Efficiency and Safety About Mild Cognitive Impairment, Randomized, Sham Device, Assessor-blinded, Multi-center Pivotal Study
Brief Title: Digital Therapeutics Research on Efficiency About Mild Cognitive Impairment Study
Acronym: DREAM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emocog Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMC-ET-101
Record Dates: First submitted 2023-06-12; First posted 2023-07-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ET-101 (Active Comparator): Treatment group
  Interventions: Device: ET-101
- Sham Device (Sham Comparator): Sham group
  Interventions: Device: Sham Device

INTERVENTIONS:
Device: ET-101 — Patients have training sessions twice a day. Each training session takes about 10~25 minutes. Cognitive training programs include meditation, cognitive training, and cognitive testing.
  Arms: ET-101
Device: Sham Device — Sham device has only cognitive function test excluding training programs.
  Arms: Sham Device

SUMMARY:
The purpose of this study is to evaluate the efficiency and safety of a digital therapeutics(ET-101) for mild cognitive impairment (MCI).

This is a randomized, sham-controlled, assessor-blinded, 24-week parallel study.

100 MCI patients will be randomly assigned to two groups. The control group will be provided with a sham device.

ELIGIBILITY:
Inclusion Criteria:

1. 55-85 years old
2. Patients diagnosed with mild cognitive impairment according to Petersen criteria

   1. A person with subjective memory complaints
   2. Memory degradation of z-score ≤ -1 from the normal range of age, gender, and level of education in the memory area of the CREAD-NP or SNSB battery
   3. The functional performance of overall cognitive function and daily life ability is sufficiently preserved.
   4. Not dementia
3. MMSE 27 or less
4. Adequate vision and hearing for clinical trial
5. Global CDR 0.5
6. If approved AD treatment drugs(AChEI, memantine, or both) are being administered, they should be administered at a stable dose for at least 12 weeks prior to randomization.
7. Have an identified trial partner (defined as someone who can assist the subject during the trial and spends at least 8 hours per week with the subject). The test partner must provide informed consent. This partner must also be willing and able to provide follow-up information to the subject during the trial. In the opinion of the investigator, the trial partner should spend sufficient time with the subject on a regular basis to ensure that the trial requirements are met. The permanent study partner does not have to live in the same residence as the subject. For study partners not residing with the subject, the investigator should ensure that the subject can easily contact the study partner while the study partner is not with the subject. If it is uncertain whether a subject's care arrangement is suitable for selection, the investigator should discuss this with the Medical Monitor. The trial partner should participate directly in visits where the clinical evaluation of CDR, EQ-5D, ADCS MCI-ADL are performed.
8. No difficulty in using mobile applications using smartphone

   1. A person who owns his/her smartphone
   2. A person who can call his/her guardian using smartphone by himself/herself
9. No difficulty in reading and writing Korean
10. Willingness and ability to comply with all aspects of the clinical trial protocol

Exclusion Criteria:

1. History of a transient ischemic attack(TIA), stroke, seizure within 12 months
2. Psychiatric symptoms that include;

   1. History of diagnosis of psychiatric disorders or symptoms that may interfere with the subject's testing procedure (e.g., psychosis, major depression)
   2. Responding "yes" to item 4 or 5 to suicidal ideation part of C-SSRS or any suicidal behavior within 6 months prior to screening, at screening or at randomization visit, or being hospitalized or treated for suicidal behavior in the past 5 years prior to screening
3. All other clinically significant abnormalities, such as

   1. Physical examinations, neurological examinations, and vital signs at screening or baseline that, in the opinion of the investigator, may require additional examination or treatment that may interfere with the study procedure or safety
   2. Other medical conditions (e.g., heart, respiratory, gastrointestinal, kidney disease) that are not adequately stable controlled or that, in the investigator's opinion, may affect the safety of the subject or interfere with the evaluation of the trial
4. A known or suspected history of drug or alcohol abuse or dependence within 2 years prior to screening
5. Prohibited concomitant medication
6. Surgery that requires general anesthesia is scheduled during the trial period.If only local anesthesia is required and the surgery is the day case without hospitalization after surgery or if, in the opinion of the investigator, the operation does not interfere with the test procedure and the safety of the subject, they should not be excluded
7. History of any type(online/offline) of cognitive intervention or participation in clinical trial regarding cognitive intervention within 12 months

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-06-08 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with the same or reduced ADAS-cog14 score | Baseline compared to month 6 (24 weeks)
  The 14 items of Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-cog14): Total scores range from 0 to 90, with higher scores indicating more worsening. Compare the proportion of subjects with the same or reduced ADAS-cog14 score between ET-101 and Sham group.

SECONDARY OUTCOMES:
Proportion of subjects with the same or reduced ADAS-cog14 score | Baseline compared to month 3 (12 weeks), month 3 compared to month 6 (12 weeks)
  ADAS-cog14: Total scores range from 0 to 90, with higher scores indicating more worsening.
Change in ADAS-cog14 total score | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  ADAS-cog14: Total scores range from 0 to 90, with higher scores indicating more worsening.
Proportion of subjects with decreased ADAS-Cog scores each at 0, 1, 2, 3, 4, 5 or more points. | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  ADAS-cog14: Total scores range from 0 to 90, with higher scores indicating more worsening.
Proportion of subjects with increased K-MMSEII score | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Korean Mini-Mental State Examination 2nd edition (K-MMSE): A score of 30 represents the least impairment and 0 represents the most severe impairment.
Change in CDR-SB | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Clinical Dementia Rating-Sum of Boxes (CDR-SB): Total scores range from 0 to 18, with higher scores indicating more worsening.
Change in K-MMSEII | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  K-MMSE II: Total scores range from 0 to 30, with lower scores indicating more worsening.
CIBIC-plus score | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Clinicians Interview-based Impression of Change (CIBIC-plus): The patient and their care giver are interviewed and questioned by the clinician. It evaluates global function and is scored from 1 (marked improvement) to 7 (marked worsening). The baseline value for CIBIC-plus is represented by Clinician's Interview-based Impression of Severity score (CIBIS).
Change in ADCOMS | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Alzheimer's Disease Composite Score (ADCOMS): Composite scores range from 0.0 to 1.97, with higher scores indicating more worsening.
Change in DSC | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Digit Symbol Coding (DSC): DSC test is sensitive to changes in information processing speed, provides measures of response speed and accuracy. A test score measures the number of correct responses in 120 seconds. A higher score indicates greater processing speed.
Change in ADCS-ADL | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  Alzheimer's Disease Cooperative Study Activities of Daily Living Inventory Scale (ADCS-ADL): Total scores range from 0 to 78, with lower scores indicating worse function.
Change in EQ-5D | Baseline compared to month 3 (12 weeks), Baseline compared to month 6 (24weeks), month 3 compared to month 6 (12 weeks)
  EuroQoL (Quality of Life)-5 Dimensions (EQ-5D): EQ-5D is a participant answered questionnaire scoring 5 dimensions - mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Total scores range from 3 (worst health state) to 1 (perfect health state).

OTHER OUTCOMES:
Adverse events rate | 12 weeks
  Adverse events rate

CONTACTS AND LOCATIONS:
Overall Officials: KeeHyung Park, Principal Investigator — Gachon University Gil Medical Center; JaeWon Jang, Principal Investigator — KangWon National University Hospital; HongJun Jeon, Principal Investigator — Konkuk University Medical Center; EoSu Kim, Principal Investigator — Severance Hospital; HyunKook Lim, Principal Investigator — Yeouido St. Mary's Hospital; YongSoo Shim, Principal Investigator — Eunpyeong St. Mary's Hospital; KeunYou Kim, Principal Investigator — SMG-SNU Boramae Medical Center
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kang S, Lim JI, Stenzel L, Kim KY, Kim E, Jeon HJ, Park DH, Lim HK, Shim Y, Jang JW, Kim Y, Lee S, Park KH. Efficacy and Safety of Mobile App-Based Metamemory Cognitive Training for Mild Cognitive Impairment: Multicenter Randomized Clinical Trial. JMIR Mhealth Uhealth. 2026 Jan 19;14:e73464. doi: 10.2196/73464. PMID 41554532